CLINICAL TRIAL: NCT02444975
Title: The Effect of Increased Water Intake on the Frequency of the Clinical Recurrent Urinary Tract Infections in Pre-menopausal Women: S-HYDRACYST
Acronym: S-HYDRACYST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NU369
Record Dates: First submitted 2015-04-29; First posted 2015-05-15 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Recurrent Urinary Tract Infection
Keywords: Urinary Tract Infections; Water intake
MeSH Terms: conditions — Urinary Tract Infections | interventions — Mineral Waters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Increased water intake+coaching program (Experimental): Women in the intervention group will be asked to increase their mineral water intake of 1.5L/day
  Interventions: Dietary Supplement: Mineral water; Other: Coaching program
- No intervention (Other): No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Dietary Supplement: Mineral water — 1.5L/day of water on top of the normal fluid intake for 1 year
  Other Names: Evian mineral water
  Arms: Increased water intake+coaching program
Other: Coaching program — Coaching program to support increased water intake
  Arms: Increased water intake+coaching program
Other: No intervention — No intervention
  Arms: No intervention

SUMMARY:
The purpose of this study is to determine whether increased water intake is effective in preventing episodes of uncomplicated urinary tract infections (UTI) in pre-menopausal women suffering from UTI recurrences.

DETAILED DESCRIPTION:
This study aims to assess the effect of increased daily water intake on the frequency of clinical, recurrent urinary tract infections (UTI) among low drinking pre-menopausal women suffering from recurrent community-acquired UTI over 12 consecutive months of study product consumption. It is a prospective, single site, open-label, randomised controlled trial in two parallel groups:

* Control group: not changing their fluid intake habits
* Intervention group: provided with mineral water, fluid intake recommendations and regular hydration coaching support

The study population consists in pre-menopausal women diagnosed with recurrent UTIs and having a 'low drinker' profile.

The total number of randomized subjects in this study is estimated at 140. The study will include only women who are low-drinkers (< 1.5 L fluids per day; urinary volume < 1.2 L per day) since they are most likely to have a predisposition to UTIs due to infrequent voiding.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 clinical recurrences of symptomatic UTI in the last 12 months
* Age ≥ 18 years

Exclusion Criteria:

* Incapacity / non-willingness to consume 1.5 L of drinking water per day on top of their usual consumption
* Women with history of UTI complications (pyelonephritis or other) in the last 12 months
* Subjects with interstitial cystitis
* Subjects with severe or uncontrolled organic disease, likely to interfere with the parameters of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2013-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Incidence of UTI | 12 months
  Difference between groups in term of UTI recurrence over 12 months of study intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Mc "Comac Medical", Sofia, Bulgaria

REFERENCES:
- [Derived] Hooton TM, Vecchio M, Iroz A, Tack I, Dornic Q, Seksek I, Lotan Y. Effect of Increased Daily Water Intake in Premenopausal Women With Recurrent Urinary Tract Infections: A Randomized Clinical Trial. JAMA Intern Med. 2018 Nov 1;178(11):1509-1515. doi: 10.1001/jamainternmed.2018.4204. PMID 30285042